CLINICAL TRIAL: NCT02626364
Title: Phase II Study of Single-agent Crenolanib in Recurrent/Refractory Glioblastoma With PDGFRA Gene Amplification
Brief Title: Study of Crenolanib in Recurrent/Refractory Glioblastoma With PDGFRA Gene Amplification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-015
Record Dates: First submitted 2015-11-03; First posted 2015-12-10 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Recurrent/Refractory Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — crenolanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): crenolanib 100mg PO TID
  Interventions: Drug: crenolanib

INTERVENTIONS:
Drug: crenolanib — single-agent crenolanib at 100 mg PO TID
  Other Names: CP-868,596-26

SUMMARY:
This is a proof of concept, single-arm study to investigate crenolanib monotherapy in patients with recurrent/refractory glioblastoma with PDGFRA gene amplification by assessing the progression-free survival (PFS) at 6 months. Crenolanib will be given orally starting at 100 mg TID continuously until disease progression, unacceptable toxicity, or consent withdrawal.

DETAILED DESCRIPTION:
This is a proof of concept, single-arm study to investigate crenolanib monotherapy in patients with recurrent/refractory glioblastoma with PDGFRA gene amplification. Eligible patients include those with recurrent/refractory glioblastoma after prior therapy including surgery, radiation, and temozolomide. The trial is designed to assess the anti-tumor activity of crenolanib in recurrent/refractory glioblastoma with PDGFRA gene amplification based on the estimation of progression-free survival (PFS) at 6 months. Symptom burden will be evaluated using the M.D. Anderson Symptom Inventory-Brain Tumor (MDASI-BT).

Crenolanib will be administered orally continuously at 100 mg TID on a 28-day cycle basis . Patients are allowed to receive crenolanib for a maximum of 26 cycles if clinical benefit has been observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) ≥ 18 years of age.
2. Histopathologically confirmed glioblastoma or gliosarcoma (WHO Grade IV) confirmed by local pathology tissue screening.
3. Radiologic evidence of first recurrence after initial treatment (including surgery, radiation, and temozolomide) or tumor refractory to initial treatment without subsequent treatment in glioblastoma or gliosarcoma (WHO Grade IV). Transformation from a lower grade glioma previously treated with radiation and/or temozolomide to glioblastoma will be considered first recurrence for the purpose of this trial
4. Tumor tissue available from original diagnosis and/or recurrence; a minimum of 1 FFPE archival tumor tissue block (preferred) or a minimum of 20 FFPE unstained slides from initial and/or most recent pre-registration biopsy or resection. It is recommended that at least 1 cm^2 of tissue composed primarily (defined as greater than 85%) of tumor is present.
5. Confirmed PDGFRA amplification in the tumor tissue at the time of diagnosis or time of recurrence. Central confirmation of PDGFRA amplification will be performed by FISH in CLIA certified lab (ProPath). Signal quantitation will be used to generate a PDGFRA/centromere 4 ratio. PDGFRA to Centromere 4 ratios will be interpreted as follows: 1.8 to 2.2, borderline for amplification; 2.2 to 5.0, low-level amplification; and greater than 5.0 or clustered signals that are too numerous to count would be considered highly amplified. Tumor samples with PDGFRA to Centromere 4 ratios of 2.2 or higher will be considered amplified and therefore eligible for this trial. For patients with local CLIA testing demonstrating PDGFRA amplification by Next Generation Sequencing (Foundation Medicine, CMS400), central testing will not be required.
6. Patients must have adequate organ function at baseline as defined below:

   • Adequate liver function (within 7 days of crenolanib commencement), as determined by:
   * Serum ALT, AST ≤ 2 × ULN
   * Normal serum total bilirubin (lower and upper limits of local Laboratory)
   * Adequate renal function assessed by: serum creatinine ≤ 1.5 × ULN
7. KPS ≥ 60
8. Recovered (returned to ≤ grade 1 as per CTCAE v4.03) from prior treatment-related toxicity.
9. A minimum of 3 weeks must have elapsed from last intake of prior standard chemotherapy treatment.
10. A minimum of 6 weeks must have elapsed from the last dose of nitrosoureas.
11. A minimum of 5 half-lives of last dose of investigational agent must have elapsed prior to C1D1.
12. More than 12 weeks from completion of chemoradiation, unless RANO criteria for early progression within 12 weeks of chemoradiation are met (See 18.1)
13. Non-pregnant and non-nursing women of childbearing potential must have a negative serum or urine pregnancy test within 3 days of crenolanib commencement ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
14. Women of childbearing potential and men must agree to use adequate contraception (simultaneous use of 2 methods of birth control) prior to study entry, for the duration of study participation and for 90 days following completion of therapy.
15. Patient able and willing to provide informed consent.
16. Ability to understand and willingness for follow-up visits.

Exclusion Criteria:

1. Pre-existing liver diseases (i.e., cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, and sclerosing cholangitis, etc.)
2. Known positive for HIV
3. Patients previously treated with bevacizumab.
4. NYHA Class III-IV heart failure, myocardial infarction <6 months prior to study entry, and/or serious arrhythmia requiring anti-arrhythmic therapy
5. Patients receiving concurrent anti-cancer treatment (chemotherapy, investigational agents, immunotherapy, endocrine therapy, or Optune®…)
6. Patients with any other severe and/or uncontrolled concurrent disease affecting the cardiovascular system, liver, kidneys, hematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures/results or compromise compliance with the protocol.
7. Pregnant or breast-feeding women.
8. Patients unable to swallow pills.
9. Patients who are allergic to MRI contrast medium or unable to undergo MRI for any other reason.
10. Patients unable to provide informed consent.
11. Patients on EIADs are not eligible, unless the antiepileptic drug can be safely tapered and discontinued before C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | 6 months

SECONDARY OUTCOMES:
Overall response rate by RANO criteria | 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 2 years
Change in symptom burden using The MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) | 2 years
Overall survival | 3 years

OTHER OUTCOMES:
Duration of response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No